CLINICAL TRIAL: NCT04414800
Title: Intranasal Ketamine Versus Intranasal Fentanyl on Pain Management in Isolated Traumatic Patients
Brief Title: Intranasal Ketamine Versus Intranasal Fentanyl
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 396828
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Multiple Trauma; Pain, Acute
MeSH Terms: conditions — Multiple Trauma; Acute Pain | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo+ Standard of Care)) (Placebo Comparator)
  Interventions: Drug: Placebo
- Ketamine + Standard of Care (Active Comparator)
  Interventions: Drug: Ketamine
- Fentanyl + Standard of Care (Active Comparator)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Placebo — Distilled water
  Arms: Control (Placebo+ Standard of Care))
Drug: Ketamine — 1 mg/kg intranasal ketamine
  Arms: Ketamine + Standard of Care
Drug: Fentanyl — 1μg/kg intranasal fentanyl
  Arms: Fentanyl + Standard of Care

SUMMARY:
Abstract Background: Given the inadequate control of pain in patients with injury that refer to the emergency departments, the rapid onset of action of intranasal administration in pain management, and the avoidance of administering opioid medications, the present study aimed at evaluating the effect of intranasal ketamine versus intranasal fentanyl on pain management in isolated traumatic patients Materials and Methods: The current study was performed on 125 patients that were divided into the following three groups: control group (n = 41), 1 mg/kg intranasal ketamine group (n = 40), and 1μg/kg intranasal fentanyl group (n = 44). Then pain scores, HR, RR, BP, and SaO2 were recorded at baseline, 5, 10, 15, 30, and 40 minutes after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute limb trauma, aged 15-65 years, with moderate to severe pain (45 mm; visual analog scale (VAS)), with a GCS score of 15, with the systolic blood pressure of lower than 180 mmHg, diastolic blood pressure of higher than 90 mmHg
* lack of pregnancy
* no history of allergy to ketamine, fentanyl (or opioids), or acetaminophen,
* no history of liver diseases,
* no acute or chronic structural or functional nasal obstruction diseases,
* no history of drug or psychiatric addiction,
* no pain medication within the past four hours,
* no history of heart disease,
* and the presentation of the written consent to participate in the study.

Exclusion Criteria:

* a decrease in GCS score to less than or equal to 14,
* an elevated systolic blood pressure to higher than 180 mmHg,
* a decreased diastolic blood pressure to less than 80 mmHg,
* inability to understand the VAS pain rating system,
* symptoms of acute heart disease and respiratory depression (respiratory rate <8 / min),
* and the patient's dissatisfaction to continue the cooperation in study

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | Change from baseline at 40 minutes
  a scale for measuring the extent of pain relief

SECONDARY OUTCOMES:
Heart rate (HR) | Change from baseline at 40 minutes
Blood pressure (BP) | Change from baseline at 40 minutes
Respiratory rate (RR) | Change from baseline at 40 minutes
SPO2 | Change from baseline at 40 minutes
  Blood oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Zahra University Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No
It will be possible to share data if requested